CLINICAL TRIAL: NCT03797560
Title: Comparison the Treatment Effects Between Ba-Duan-Jin and Pregabalin in Patients with Fibromyalgia
Brief Title: Comparison of Ba-Duan-Jin and Pregabalin in Patients with Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Juan Jiao, Deputy chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z181100001718153
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Eight Brocades; Ba-Duan-Jin; Baduanjin; Qigong; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ba-Duan-Jin group (Experimental): Ba-Duan-Jin therapy: The participants will be guided by a research staff to do the Ba-Duan-Jin therapy for 50 minutes twice weekly for 12 weeks, in the outpatient section of the hospital.
  Placebo pregabalin capsules: Pregabalin placebo treatment will be administered at bedtime once a day, starting at 150 mg for the first week, and increase to the dose of 300 mg from the second week. After one week, if 300 mg dose is tolerable, then maintain it for 10 additional weeks, if not, then go back to the 150 mg dose for 10 additional weeks.
  Interventions: Other: Ba-Duan-Jin
- Pregabalin group (Active Comparator): Wellness education and muscle relaxation exercise program: This program will be held for 50 minutes twice weekly for twelve weeks, containing 10-minute wellness education, 10-minute doctor-patient discussion, and 30-minute guided muscle relaxation exercise.
  Active pregabalin capsules: As same usage as the placebo pregabalin capsules.
  Interventions: Drug: Pregabalin capsule

INTERVENTIONS:
Other: Ba-Duan-Jin — Ba-Duan-Jin is a common form of "self-health-care" Qigong exercise that has been practiced by Chinese people for at least eight hundred years. It consists of eight sets of simple movements. By combining meditation with slow, graceful movements, deep breathing, and relaxation, Ba-Duan-Jin practitioners believe it has the ability to move vital energy (Qi) throughout the body. Ba-Duan-Jin is also considered to be a multicomponent intervention that integrates physical, psychosocial, emotional, spiritual, and behavioral elements. While the biological mechanisms remain unclear, previous clinical trials have demonstrated that Ba-Duan-Jin can improve sleep quality, physical health, and mental health in patients with various chronic diseases
  Other Names: Baduanjin; Eight Brocades; Eight-Section Brocade
  Arms: Ba-Duan-Jin group
Drug: Pregabalin capsule — Pregabalin is one of the three medications (pregabalin, duloxetine, and milnacipran) that have been approved by the Food and Drug Administration (FDA) to treat fibromyalgia in US, and the only medicine that has been approved in China.
  Arms: Pregabalin group

SUMMARY:
Fibromyalgia is a chronic debilitating musculoskeletal pain syndrome. Pregabalin is the only medication that has been approved to treat fibromyalgia in China. Currently, there has been a growing interest in the development of non-pharmacological therapies. Ba-Duan-Jin is an ancient Chinese exercise for health promotion yet easy to learn. Findings from our previous study showed an effectiveness and good safety of Ba-Duan-Jin in patients with fibromyalgia. This study is to evaluate the effectiveness comparison of Ba-Duan-Jin and pregabalin in managing fibromyalgia symptoms experienced by Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* meet the 1990 American College of Rheumatology (ACR) Research Classification Criteria for fibromyalgia;
* be between the ages of 18 to 70 years.

Exclusion Criteria:

* had practiced Ba-Duan-Jin, Tai Chi, yoga or other forms of Qigong exercise within 12 months of their recruitment to the study;
* be less than 40mm of pain VAS score;
* had renal failure, and severe depression or anxiety;
* had any poorly-controlled comorbid medical conditions, such as dementia, cancer, thyroid disease, inflammatory arthritis;
* pregnancy or planned pregnancy within the study period;
* patients residing more than 70 miles from the research site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The change of the Visual Analogue Scale (VAS) for pain from baseline. | up to 1 week
  Pain VAS, range, 0 to 100 mm, where higher scores indicated the perceived pain to be more severe.

SECONDARY OUTCOMES:
The change of the revised Fibromyalgia Impact Questionnaire (FIQR) from baseline. | Baseline, week 4, week 8, and week 12.
  A self-administered questionnaire with 10 subscales, measuring fibromyalgia symptoms and function domains. FIQR total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
The change of the Multidimensional Fatigue Inventory-20 (MFI-20) from baseline. | Baseline, week 4, week 8, and week 12.
  The Multidimensional Fatigue Inventory-20 (MFI-20) measures fatigue severity. The MFI-20 total score ranges from 0 to 80, with higher scores indicate more severe fatigue.
The change of the Pittsburgh Sleep Quality Index (PSQI) from baseline. | Baseline, week 4, week 8, and week 12.
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.
The Beck II Depression Inventory (BDI) | Baseline, week 4, week 8, and week 12.
  The Beck II Depression Inventory (BDI) assesses the severity of depressive symptoms. Scores range from 0 to 39, with higher scores indicate a greater degree of depression severity.
The change of the Perceived Stress Scale (PSS) from baseline. | Baseline, week 4, week 8, and week 12.
  The Perceived Stress Scale (PSS) is for measuring the perception of stress and current levels of experienced stress. Scores range from 0 to 56, with higher total score indicating a greater degree of symptom severity.
Global Impression of Change (PGIC) questionnaire evaluated at week 12. | Week 12.
  A questionnaire determine any change in overall symptom status from the beginning of the study to its conclusion (score range, 1 [very much improved] to 7 [very much worse).
The change of the Short Form-36 Health Status Questionnaire (SF-36) from baseline. | Baseline, week 4, week 8, and week 12.
  The Short Form-36 Health Status Questionnaire (SF-36), which measured health-related quality of life (range, 0 to 100, with higher scores indicating better perceived health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiao Juan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Li YT, Sun YR, Wang J, Li Y, Zhang JH, Jiao J, Jiang Q. Therapeutic Effects of Ba-Duan-Jin versus Pregabalin for Fibromyalgia Treatment: Protocol for a Randomized Controlled Trial. Rheumatol Ther. 2021 Sep;8(3):1451-1462. doi: 10.1007/s40744-021-00341-9. Epub 2021 Jul 22. PMID 34292537
- See also: In this article the study protocol and background are described — https://doi.org/10.1007/s40744-021-00341-9